CLINICAL TRIAL: NCT05923762
Title: Oral Health Related Quality of Life and Its Implications for Dental Health Care - a Swedish National Survey
Brief Title: Oral Health Related Quality of Life
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dalarna County Council, Sweden (Other)
Collaborators: Region Gävleborg (Other)
Responsible Party: Principal Investigator, Kristina Edman, Principal Investigator, Dalarna County Council, Sweden
Other Study IDs: OHRQoL
Record Dates: First submitted 2023-06-15; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Oral Health Related Quality of Life; Oral Disease
MeSH Terms: conditions — Mouth Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 18-85 years of age
  Interventions: Behavioral: OHRQoL

INTERVENTIONS:
Behavioral: OHRQoL — Oral health-related quality of life will be measured by the "Oral Impact on Daily Performance" (OIDP)

SUMMARY:
As oral health has a major impact on general health and quality of life, good oral health are essential. The aspects of oral health that are most important for each individual vary, and quality of life is subjective, and influenced by the person´s experiences, perceptions, expectations and ability to adapt to circumstances. FDI World Dental federations definition of oral health is; "Oral health is multifaceted and includes the ability to speak, smile, smell, taste, touch, chew, swallow, and convey a range of emotions through facial expressions with confidence and without pain, discomfort, and disease of the craniofacial complex.

ELIGIBILITY:
Inclusion Criteria: Read and understand Swedish -

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The target population is adults aged 18-85 years that resides in Region Dalarna, Sweden.
Sampling Method: Probability Sample
Enrollment: 3700 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
OHRQoL | 2024-01-15 - 2024-12-31
  Questionnaire, Oral health problems in the last six months with eating, cleaning teeth, socializing. The questionnaire used will be OIDP